CLINICAL TRIAL: NCT05617638
Title: Impact of Virtual Reality (e-Nature VR) During Hospitalization in Adult Intensive Care Unit
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was definitively suspended due to the difficulty in including participants to reach the appropriate sample size
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Beneficência Portuguesa de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: e-Nature VR - ICU
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2024-09

CONDITIONS: Pain
Keywords: virtual reality; intensive care unit; nature; wellness
MeSH Terms: conditions — Pain | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (No Intervention): The control group will not have access to VR.
- Intervention Group (Active Comparator): Participants in the intervention group will use VR for 20 minutes for 2 consecutive days.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Participants will watch nature images in virtual reality from the e-Natureza VR Database for 20 minutes for 2 consecutive days.
  Other Names: e-Nature VR
  Arms: Intervention Group

SUMMARY:
Randomized clinical trial to analyze the perceived impact of the virtual reality intervention on the experience of pain and well-being, and the influence on vital signs and the relationship with the length of stay in the intensive care unit.

DETAILED DESCRIPTION:
The highly specialized and complex technology used in intensive care units to provide continuous monitoring of the patient health context makes possible to increase the survival of patients with critical and unstable clinical status, but increases the triggering factors of the stress of hospitalized patients. Staying in these therapy units is accompanied by additional stress, confusional mental states, cognitive dysfunction, and depression. Virtual reality is a technique that involves the use of computer technology to create the effect of an interactive three-dimensional world in which objects have a spatial presence reducing the suffering related to a medical procedure, without side effects and without the need for additional personnel. Actual exposure to nature can be difficult to achieve for patients admitted to intensive care. Therefore, exposure to nature via media devices, and virtual reality (VR) is considered a promising technology due to its advantage in creating a sense of immersion. Furthermore, some evidence indicates that virtual nature can improve attentional resources, cognitive performance, and pain experience.

This clinical trial aims to analyze the influence of VR use in patients of Intensive Care Unit (ICU). After informed the consent form, participants will be randomly into control and intervention groups. Blood pressure, heart rate, respiratory rate, oxygen saturation will be evaluated, in addition to the experience of well-being and pain immediately before and immediately after the intervention for 2 consecutive days.The hypothesis of the study is that VR will positively influence vital signs and lived experiences, which will consequently reduce the length of stay in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* individuals of both sexes;
* without communication, vision, hearing or intellectual disabilities;
* capable of mental to fill in the questionnaires;
* who watch at least 5 minutes of the video, minimum physiological immersion time.

Exclusion Criteria:

* use of sedatives;
* those who experience considerable discomfort possibly caused by virtual reality such as nausea, dizziness or headache, with a history of vertigo, nausea, vomiting;
* convulsion, labyrinthitis, epilepsy, dementia, mental confusion, psychomotor agitation;
* claustrophobia or expressing a desire to discontinue the study;
* patients who use anticholinergic drugs (antipsychotics and benzodiazepines);
* delirium;
* clinical worsening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2023-06-27 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Oxygen Saturation Percentage at post intervention. | Immediately post-intervention for 2 consecutive days.
  Quantify the change from baseline of pulse oximetry on the monitor in the intensive care unit, immediately after the intervention on the first day of Virtual Reality use (D1) and immediately after on the second day (D2).
Change from Baseline Blood Pressure Values at post intervention. | Immediately post-intervention for 2 consecutive days.
  Quantify the change from baseline of blood pressure values on the monitor in the intensive care unit, immediately after the intervention on the first day of Virtual Reality use (D1) and immediately after on the second day (D2).
Change from Baseline Respiratory Rate Values at pos intervention. | Immediately post-intervention for 2 consecutive days.
  Quantify the change from baseline of respiratory rate values on the monitor in the intensive care unit, immediately after the intervention on the first day of Virtual Reality use (D1) and immediately after on the second day (D2).
Change from Baseline Heart Rate Values at pos intervention. | Immediately post-intervention for 2 consecutive days.
  Quantify the change from baseline of heart values on the monitor in the intensive care unit, immediately after the intervention on the first day of Virtual Reality use (D1) and immediately after on the second day (D2).
Change from Baseline Pain Perception at pos intervention. | Immediately post-intervention for 2 consecutive days.
  Will be applied the Visual Analogue Scale - VAS. It is one of the most used instruments for pain assessment with a score from 0 to 10 that allows the patient to evaluate the pain of the procedure through a visual analogue scale numbered from zero to ten, with zero no pain, ten being the worst pain ever felt in life.The scale will be applied immediately after the first day (D1) of intervention using Virtual Reality and immediately after the second day (D2).
Change from Baseline Affective States pos intervention. | Immediately post-intervention for 2 consecutive days.
  Will be applied the Positive and Negative Affect Schedule - PANAS. It is one of the most used instruments in the investigation of affective states composed of 20 questions and each item can be rated on a likert type frequency scale of sensations, raging from 0 (not at all) to 5 (extremely). The questionnaire will be applied immediately after the first day (D1) of intervention using Virtual Reality and immediately after the second day (D2).

SECONDARY OUTCOMES:
Change in length of stay in the intensive care unit pos intervention | Immediately post-intervention for 2 consecutive days.
  The days of hospitalization in intensive care of patients in the intervention group will be evaluated and will be compared with the days of stay in the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Eliseth R Leão, PhD, Principal Investigator — Hospital Israelita Albert Einstein; Roberta M Savieto, MNP, Study Chair — Hospital Israelita Albert Einstein; Gabriela AG Gouveia, BPT, Study Chair — Beneficência Portuguesa de São Paulo
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rousseaux F, Dardenne N, Massion PB, Ledoux D, Bicego A, Donneau AF, Faymonville ME, Nyssen AS, Vanhaudenhuyse A. Virtual reality and hypnosis for anxiety and pain management in intensive care units: A prospective randomised trial among cardiac surgery patients. Eur J Anaesthesiol. 2022 Jan 1;39(1):58-66. doi: 10.1097/EJA.0000000000001633. PMID 34783683